CLINICAL TRIAL: NCT07026825
Title: Surgical Resection Improves Survival in Gastric-type Endocervical Adenocarcinoma: A SEER-Based Propensity-Matched Cohort Study
Brief Title: Surgical Resection Enhances Survival in Gastric-type Endocervical Adenocarcinoma: A SEER-Based Study
Acronym: SURGE
Status: Completed | Type: Observational
Sponsor: Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other)
Responsible Party: Sponsor
Other Study IDs: JS2024-32-1
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Gastric-type Endocervical Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgical Resection Group: Participants in this group undergo standard surgical resection aimed at the complete or partial removal of tumor tissue. The type of surgery-open or minimally invasive-is determined based on the patient's clinical condition and the surgeon's judgment. Preoperative and/or postoperative adjuvant therapies, such as chemotherapy or radiotherapy, may be administered to enhance treatment efficacy.
- Non-Surgical Management Group: Participants in this group receive standard non-surgical treatments, including chemotherapy, radiotherapy, targeted therapy, or immunotherapy. The specific treatment regimen is tailored to the patient's condition and determined by the treating physician, aiming to control tumor progression, alleviate symptoms, and improve quality of life.

SUMMARY:
This retrospective cohort study analyzes the effect of surgical resection on survival outcomes in patients with gastric-type endocervical adenocarcinoma (GAS), using data from the SEER database (2000-2021). Propensity score matching and multivariable Cox regression were used to compare overall survival (OS) and tumor-specific survival (TSS) between patients who underwent surgery and those who did not. The study aims to determine whether primary tumor resection is associated with improved survival across tumor sizes and stages.

DETAILED DESCRIPTION:
The study utilized de-identified data from the SEER program encompassing women aged ≥18 with histologically confirmed gastric-type endocervical adenocarcinoma between 2000 and 2021. The primary endpoints were overall survival and tumor-specific survival. Statistical analyses included multivariable Cox regression, propensity score matching (2:1), and inverse probability of treatment weighting (IPTW). Subgroup analyses were performed based on FIGO stage and tumor size (>4 cm). A total of 308 eligible cases were included. No patient interaction or clinical intervention occurred.

ELIGIBILITY:
Inclusion Criteria:

Histologically confirmed gastric-type endocervical adenocarcinoma Cervix as the first primary site Diagnosis between 2000 and 2021

Exclusion Criteria:

Incomplete survival or treatment data Diagnosis not confirmed microscopically

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients aged 18 years and older with histologically confirmed gastric-type endocervical adenocarcinoma and no prior history of other malignancies.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Outcome | Time from diagnosis to death from any cause Up to 22 years (2000-2022)
  Overall Survival (OS)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to concerns regarding participant privacy and confidentiality, as well as the absence of participant consent for data sharing.